# **PROTOCOL**

# Selective Coronary Revascularization in Peripheral Artery Disease patients after lower-extremity revascularization (SCOREPAD trial)

Working draft protocol version number: Latvia RCT/PAD/15012024

Universal Trial Number: TBA

In the following, Institute of Science, Pauls Stradins clinical university hospital and its affiliates will be stated as "Stradins university hospital".

This confidential document is the property of Stradins university hospital. No unpublished information contained herein may be disclosed without prior written approval from Stradins university hospital. Access to this document must be restricted to relevant parties.

| DOCUMENT HISTORY | | |
|---|---|---|
| Document version | Date | Applicable in country(-ies) and/or site(s) |
| 1.0 | 21 January 2024 | All |

**Study Objective** To determine whether the diagnosis of ischemia-producing coronary

stenosis together with selective coronary revascularization in PAD patients following lower-extremity revascularization can reduce adverse

cardiac events and improve survival compared to PAD patients

receiving standard cardiac evaluation and treatment.

Study Design Multicenter, prospective randomized clinical trial of patients with stable

PAD and no known CAD who had undergone open or endovascular lower-extremity revascularization for CLTI or severe claudication. Eligible patients will be randomly assigned to receive (a) current guideline-directed care with evidence-based best medical therapy

(BMT) and risk factor control or (b) in addition to BMT and risk factor


control, non-invasive cardiac evaluation using coronary CTA and FFRct to identify ischemia-producing coronary lesions together with selective ischemia-targeted coronary revascularization. The primary outcome measure will be MACE (myocardial infarction, urgent coronary revascularisation, cardiac death) during 2 years follow up with secondary endpoints of myocardial infarction, cardiac death, urgent coronary revascularisation, all-cause death.

Principal Investigator:

Dainis Krievins, MD, PhD and principal Co-investigator Andrejs Erglis MD, PhD

Pauls Stradins Clinical University hospital

13 Pilsonu street

Riga, Latvia. LV-1002

Dainis.krievins@gmail.com; dainis.krievins@stradini.lv

+371 29450000; +371 67069604

Co-investigators & Steering committee: Christopher K. Zarins MD; Marianne Brodmann MD, PhD; Gustavs Latkovskis MD, PhD; Indulis Kumsars MD, PhD; Peteris Stradins MD, PhD; Sanda Jegere MD, PhD; Patricija Ivanova MD, PhD and others TBA.

**Study Sites:** Pauls Stradins Clinical University Hospital plus up to 10 additional sites

**CRO:** Institute of Science, Pauls Stradins Clinical University Hospital

**Study Sponsor:** Pauls Stradins Clinical University Hospital with a grant from the

Latvian Council of Science Nr. VPP-VM-Veseliba-2023/3-0004.


## I. BACKGROUND

Patients with symptomatic peripheral artery disease (PAD) are at high risk for adverse cardiac events and have poor long-term survival due to coexistent coronary artery disease (CAD). The risk of death is particularly high for patients with critical limb threatening ischemia (CLTI) with 20% one-year and 60% five-year mortality.<sup>2,3</sup> This mortality rate is higher than for symptomatic CAD and most cancers.<sup>4</sup> Moreover, this high mortality rate has remained unchanged over the past 40 years despite remarkable advances in medical treatment and interventional therapies.<sup>5</sup> In the randomized BASIL (Bypass Versus Angioplasty in Severe Ischaemia of the Leg) trial, which was conducted 20 years ago, all-cause mortality in both groups was 56% at 5 years. In a recent review of 168.553 Medicare beneficiaries revascularized with current endovascular techniques the 5-year mortality rate was 55%. Most recently the US based BEST-CLI trial and the European based BASIL-2 trial both reported 50% 5-year mortality in both arms of the study regardless of whether LE revascularization was using open or endovascular techniques. While it well known that most PAD patients have significant CAD and that symptomatic PAD is a powerful independent predictor of cardiovascular death, guidelines do not recommend preoperative cardiac testing, particularly in patients without cardiac symptoms, due to lack of evidence that coronary revascularization improves long-term outcome.8 Rather, efforts to improve the survival of PAD patients have been focused on optimizing medical treatment and aggressive risk factor control to limit the progression of systemic atherosclerosis. While medical therapy has reduced mortality in large CAD trials that include patients with PAD<sup>10</sup>, there is no evidence that best medical therapy has improved the survival PAD patients following lower-extremity revascularization.<sup>5,11-13</sup>

The potential benefit of coronary revascularization to improve the survival of PAD patients was first brought to light by Hertzer, et al. in a landmark study of 1000 coronary angiograms in vascular surgery patients 4 decades ago. However, this strategy fell by the wayside due to lack of randomized trial evidence showing that coronary revascularization improved long-term survival of PAD patients. The most recent trial, the Coronary Artery Revascularization Prophylaxis (CARP) trial was conducted two decades ago using angiography-guided coronary revascularization rather than the current standard of fractional flow reserve (FFR)-guided revascularization which has been shown to reduce mortality. Furthermore, the requirement for pre-operative coronary revascularization in CARP resulted in a two-month delay of the vascular surgery procedure, which is not an option for most CLTI patients. The alternative strategy of coronary revascularization after peripheral revascularization in order to reduce adverse coronary events and improve long-term survival has not been evaluated in controlled clinical trials. This may be due to lack of a reliable non-invasive method for identifying PAD patients with occult hemodynamically significant coronary stenosis who may benefit from coronary revascularization.


A new non-invasive cardiac diagnostic test, coronary CT-derived fractional flow reserve (FFR<sub>CT</sub>) provides a unified anatomic and functional assessment of coronary artery disease which can reliably identify ischemia-producing coronary lesions.<sup>18</sup> FFR<sub>CT</sub> accurately reflects invasively measured FFR and can help guide patient management and coronary revascularization decisions.<sup>19,20</sup> In a single center study, of CLTI patients with no known CAD who were scheduled for lower-extremity revascularization, systematic pre-operative FFR<sub>CT</sub> evaluation revealed a high prevalence (69%) of unsuspected (silent) ischemia-producing coronary stenosis (FFR<sub>CT</sub> ≤0.80).<sup>21</sup> While this did not result in postponement of the revascularization procedure, it identified high-risk patients and facilitated multidisciplinary vascular team care, including selective coronary revascularization of high-risk coronary lesions following recovery from lower-extremity revascularization.<sup>22</sup> This resulted in improved one, two and 3-year survival of PAD patients compared to control patients receiving guideline-directed cardiac evaluation and care.<sup>22,23</sup> The purpose of this study is to determine whether FFR<sub>CT</sub>-guided coronary revascularization of PAD patients with asymptomatic (silent) coronary ischemia after recovery from lower-extremity revascularization can reduce adverse cardiac events and improve survival compared to PAD patients with no coronary symptoms receiving standard cardiac evaluation and care.

## II. OBJECTIVE

The primary objective of this study is to determine whether among symptomatic PAD patients with no known CAD who had undergone lower-extremity revascularization, a strategy of best medical therapy (BMT) plus selective coronary revascularization based on FFRct assessment of lesion-specific coronary ischemia can reduce adverse cardiac events and improve survival compared to BMT alone. Lesion-specific coronary ischemia is defined as  $FFR_{CT} \le 0.80$  distal to stenosis in a major ( $\ge 2$  mm) coronary artery with severe ischemia defined as  $FFR_{CT} \le 0.75$ .

## III. STUDY ENDPOINTS

The primary endpoint of the study is a composite of cardiac death, myocardial infarction (MI) or urgent coronary revascularisation (MACE) during 2 years follow up. Secondary endpoints include MI, cardiac death, urgent coronary revascularisation, cardiovascular (CV) death, all-cause death during follow up.

## IV. STUDY DESIGN

This study targets a population of patients with symptomatic PAD (CLTI or severe claudication in 1:1 ratio) and no prior cardiac history, no myocardial infarction, no coronary angiography or coronary CTA, and no coronary revascularization (PCI or CABG) who have undergone successful lower extremity revascularization with planned post-operative best medical therapy. Within 14 days following lower-extremity revascularization, patients will be randomly assigned to BMT alone or BMT plus coronary CT angiography (which must be completed within 14 days of randomization) and FFRct analysis to determine the functional significance of coronary lesions identified on the CT scan. Results of the CT scan and


FFR<sub>CT</sub> analysis in patients randomized to the CT-FFRct group, will be provided to treating physicians to help guide patient management with Heart Team consideration for coronary angiography and revascularization as appropriate for each patient. Coronary revascularisation (PCI or CABG), if indicated, is strongly reccomended within 3 months from the randomisation. Clinical follow up (based on date of randomization) is planned 6 months, one and 2 years. Additional long-term follow up out to 5-years is planned for participating centers. An independent academic clinical events committee will adjudicate all endpoints in a blinded manner. The definition of outcome events will be in accordance with Academic Research Consortium-2 consensus document<sup>26</sup>. Sample size power calculations assumed a hazard ratio of 0.5 with estimated sample size up to 600 patients (up to 300 in each group), 90% power, alpha .05. The patient sample size may be reduced if statistical significance been achieved.

## V. INCLUSION AND EXCLUSION CRITERIA

## **Inclusion Criteria**

- 1. Inform consent obtained before any study-related activities
- 2. Age above or equal to 50 years with symptomatic lower extremity PAD (severe claudication or chronic limb-threatening ischemia, Rutherford 3,4,5) which has been successfully revascularized by open surgical or endovascular procedure within the past 14 days
- 3. Willing and able to undergo coronary CTA scan within 14 days of randomization and agrees to submission of CTA data set for HeartFlow FFRct analysis with results made available to treating physician

## **Exclusion Criteria**

- 1. Known CAD, history of MI, prior coronary revascularization (PCI or CABG)
- 2. Patient underwent coronary angiography or coronary CTA before the randomization
- 3. Known hystory of 2<sup>nd</sup> or 3<sup>rd</sup> degree heart block; sick sinus syndrome; long QT syndrome
- 4. History of severe asthma, severe or bronchodilator-dependent COPD
- 5. Severe congestive heart failure (NYHA III or IV)
- 6. Severe arrhythmia, prior pacemaker or internal defibrillator lead implantation
- 7. Impaired chronic renal function (EPI-GFR<30ml/min)
- 8. Subjects with known anaphylactic allergy to iodinated contrast
- 9. Pregnancy or unknown pregnancy status in subject of childbearing potential
- 10. Evidence of ongoing or active clinical instability, including acute chest pain (sudden onset), cardiogenic shock, unstable blood pressure with systolic blood pressure <90 mmHg, or acute pulmonary edema


- 11. Any active, serious, life-threatening disease with a life expectancy of less than 2 years
- 12. Any active infection
- 13. Inability to comply with study procedures
- 14. Contraindication for guideline-guided longterm antiplatelet/anticoagulation regime after PCI/CABG
- 15. Participation in any interventional clinical study within 30 days prior to screening

# VI. Rules for subject withdrawal and terminating the study

In accordance with the Declaration of Helsinki, as amended, each subject is free to withdraw from the study at any time. Investigator(s) also have the right to withdraw subjects from the study in the event of illness, adverse events (AEs), serious adverse events (SAEs), other reasons concerning the health or well being of the subject, or in the case of lack of cooperation. The reason for withdrawal must be noted in the Case Report Forms (CRFs). If the reason for withdrawal is a clinical AE or SAE, follow up of the subject will continue until the outcome is evident. The specific event or test result(s) must be recorded in the CRFs.

There are no formal termination criteria for this study. The sponsor reserves the right to terminate the study at any time. Investigators have the responsibility to comply with International Conference on Harmonization E6-Good Clinical Practice (ICH E6 - GCP) guidance. The sponsor, the IRB, or the health authorities may terminate a center for the following (but not limited to) reasons:

- 1) Failure of the investigator to comply with pertinent E6-GCP guidelines and regulations
- 2) Serious protocol violations
- 3) Submission of knowingly false information from the research facility.

## VII. Ethical Considerations

The potential benefits to all subjects participating in this study is that they may receive closer monitoring and follow up with better compliance to guideline-recommended BMT and risk factor control. Patients randomized to the coronary CTA-FFRct arm of the study will have additional benefit of specific cardiac diagnosis and treatment. Prior studies have demonstrated that PAD patients often have unrecognized coronary artery disease and that they have a high risk of cardiovascular complications including MI and cardiovascular death. Current guideline-directed pre-procedure cardiac evaluation of PAD patients without cardiac symptoms does not include cardiac imaging or stress testing. Half of enrolled subjects within the study will undergo coronary artery CT scanning which is highly sensitive for detecting CAD. Subsequent FFRct analysis will identify those with hemodynamically significant coronary stenosis. The incremental potential risks to subjects participating in the study are solely and directly related to the performance of the additional cardiac diagnostic testing in half of the patients.


# VIII.A. Risks of Coronary CTA

Coronary CTAs expose subjects to small amounts of ionizing radiation. Since the introduction of 64-detector row CTA scanners in 2005, numerous radiation dose reduction methods have been developed which now permit CTA performance with low overall radiation dose. Minimization of radiation dose while preserving image quality is a goal of the study; optimization of radiation dose may be achieved by a by a combination of 7 additive dose reduction strategies: ECG dose modulation; Weight-based tube voltage; Prospective ECG triggering; Minimization of "padding"; Minimization of Z-axis coverage; Limiting of the field of view (FOV); Automatic exposure control. Coronary CTA performance necessitates the use of iodinated contrast. Minor reactions to x-ray contrast material can occur, including itches or hives with an incidence of approximately 1 in 200 subjects. More severe reactions that are very infrequent include hypotension, laryngospasm and bronchospasm. The incidence of these reactions is estimated at about 1 in 5,000 and is treated with intravenous epinephrine. Extravasation of x-ray contrast material outside the vein during injection may occur and result in a painful soft tissue swelling and bruising. Subjects will be monitored for extravasation during injection and the amount of contrast material injected into the tissues is usually quite small without significant clinical consequences.

# VIII.B. Risks of FFRCT analysis

In subjects with Coronary CTA, FFR<sub>CT</sub> analysis will be performed using the clinically acquired Coronary CTA data set. The FFR<sub>CT</sub> analysis in these subjects does not require additional imaging. There is no additional risk to the subject.

# IX. STUDY PROTOCOL REQUIREMENTS

- 1. After providing informed consent, each subject will undergo the following assessments as indicated on CRF:
  - a. Collection of demographic information, including height and weight
  - b. A summary of index PAD revascularization procedure
  - c. A summary of the subject's relevant medical and surgical history (Diabetes mellitus, Dyslipidemia, Arterial hypertension, Smoking)
  - d. Recording of concurrent and concomitant medications

## 2. Coronary CTA (cCTA) Procedure

- 1) Perform cCTA with strict adherence to SCCT guidelines including, but not limited to:
  - a. Heart rate control: administration of  $\beta$ -blockers, if needed, to achieve a heart rate of <60 bpm
  - b. CT image acquisition after administration of sublingual nitrate spray or after administration of sublingual nitrate tablet (3-5 minutes)


- c. using breath-holding and other techniques to minimize motion artifact
- d. contrast protocols: bi-phasic injection protocol
- e. kV/mA settings per ALARA principles. Patients who weigh more than 70kg should be scanned at 120kV.
- 2) The additional thorax CT findings (pulmonaly oncology, etc.) might be collected at selected sites.
- 3. Post-procedure follow up data from clinical visits and/or phone calls 6 months, one and 2 years (annually up to 5 years for patients entering prolonged study at participating sites).
- 4. Open label randomization will be done after patient screening at approximate rate 1:1 CLTI to claudicants (Rutherford III,IV).

# X. Case Report Forms

Electronic or paper case report forms will used.

## XI. Institutional Review

Before starting this study, the protocol will be submitted to the regulatory bodies/local health authorities (in accordance with local regulations) and the study will not start before the EC/IRB gives written approval or a favorable opinion in accordance with ICH E6-GCP and all applicable regulatory bodies/local health authorities give approval or a favorable opinion as required.

## XII. Informed consent

Written and oral information about the study in a language understandable by the subject will be given to all subjects by the investigator and/or designee. The subject's willingness to participate in the study will be documented in writing in a consent form, which will be signed by the subject with the date of that signature indicated. The investigators will keep the original consent forms and copies will be given to the subjects. The informed consent will also be signed and dated by the person who conducted the informed consent discussion.

## XIII Confidentiality regarding study subjects

The investigator(s) must assure that the privacy of the subjects, including their personal identity and all other personal medical information, will be maintained at all times. In documents or image material submitted to the sponsor, subjects will not be identified by their names, but by an identification code. Personal medical information may be scrutinized for the purpose of verifying data recorded in the CRF. This may be done by properly authorized persons, the quality assurance unit, or regulatory authorities. Personal medical information will always be treated as confidential.


#### **XIV Financial Disclosure**

The investigator(s) (or investigating institution) will provide the sponsor with accurate financial disclosure regarding real or potential financial conflicts of interest.

## XV Insurance

As there is no any invasive investigation product been tested, the local site clinical liability insurance will be in power to cover malpractice.

## XVI Adverse event and serious adverse event reporting

Only endpoints and adverse events (AE) listed in amendment should be repoted according to ICH-GCP requrements. A Clinical Adjudication committee will evaluate all Study Endpoints.

## REFERENCES

- 1. Golomb BA, Dang TT, Criqui MH. Peripheral arterial disease: morbidity and mortality implications. Circulation 2006;114:688-699.
- 2. Mustapha JA, Katzen BT, Neville RF, et al. Disease burden and clinical outcomes following initial diagnosis of critical limb ischemia in the Medicare population. JACC Cardiovasc Interv. 2018;11:1011-12.
- 3. Baubeta Fridh, E, Andersson M, Thuresson M, Sigvant, B, Kragsterman, B, Johansson S, et al. Amputation rates, mortality, and pre-operative comorbidities in patients revascularised for intermittent claudication or critical limb ischemia: a population based study. Eur J Vasc Endovasc Surg 2017;54:480-6.
- 4. Teraa M, Conte MS, Moll FL, Verhaar MS. Critical limb ischemia: current trends and future directions. J Am Heart Assoc 2016;5:e002938.
- 5. Sigvant B, Kragsterman B, Falkenberg M, Hasvold P, Johansson S, Thuresson M, et al. Contemporary cardiovascular risk and secondary prevention drug treatment patterns in peripheral artery disease patients undergoing revascularization. J Vasc Surg 2016;64:1009-17.
- 6. Bradbury AW, Adam DJ, Bell J, Forbes JF, Fowkes GR, Gillespie I, et al. Bypass versus Angioplasty in Severe Ischaemia of the Leg (BASIL) trial: an intention-to-treat analysis of amputation-free and overall survival in patients randomized to a bypass surgery-first or a balloon angioplasty-first revascularization strategy. J Vasc Surg 2010;51:5S-17S.
- 7. Secemsky EA, Shen C, Schermerhorn M, Yeh RW. Longitudinal assessment of safety of femoropopliteal endovascular treatment with paclitaxel-coated devices among Medicare beneficiaries: the SAFE-PAD study. JAMA Intern Med 2021;doi:10.1001/jamainternmed.2021.2738.


- 8. Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, et al. 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg 2018;55:305-68.
- 9. Conte MS, Bradbury AW, Kolh P, White JV, Dick F, Fitridge R, et al. Global vascular guidelines on the management of chronic limb-threatening ischemia. J Vasc Surg 2019;69:3S-125S.
- 10. EikelboomJW, Bhatt DL, Foxx KAA, Bosche J, Connolly SJ, Anand S, et al. Mortality benefit of rivaroxaban plus aspirin in patients with chronic coronary or peripheral artery disease. J Am Coll Cardiol 2021;78:14-23.
- 11. Thiney M, Schiava ND, Ecochard R, Feugier P, Lermusiaux P, Millon A, et al. Effect on mortality and cardiovascular events of adherence to guideline-recommended therapy 4 years after lower extremity arterial revascularization. Ann Vasc Surg 2018;52:138-46.
- 12. Bonaca MP, Nault P, Giugliano RP, Keech AC, Pineda AL, Kanevsky E, et al. Low-density lipoprotein cholesterol lowering with evolocumab and outcomes in patients with peripheral artery disease: insights from the FOURIER trial. Circulation 2018;137:338-350.
- 13. Bonaca MP, Bauersachs RM, Anand SS, Debus ES, Nehler MR, Patel MR et al. Rivaroxaban in peripheral artery disease after revascularization. N Engl J Med 2020;383:2089-2090.
- 14. Hertzer NR, Beven EG, Young JR, O'Hara PJ, Ruschhaupt WF, Graor RA, et al. Coronary artery disease in peripheral vascular patients: a classification of 1000 coronary angiograms and results of surgical management. Ann Surg 1984;199:223-33.
- 15. McFalls EO, Ward HB, Moritz TE, Goldman S, Krupski WC, Littooy F, et al. Coronary-Artery Revascularization before Elective Major Vascular Surgery. N Engl J Med 2004;351:2795-804.
- 16. Xaplanteris P, Fournier S, Pijls NHJ, Fearon WF, Barbato E, Tonino PAL, et al. Five-Year Outcomes with PCI Guided by Fractional 383 Flow Reserve. N Engl J Med 2018;379:250-259.
- 17. Volz S, Dworeck C, Redfors B, Petursson P, Angeras O, Gan LM, et al. Survival of patients with angina pectoris undergoing percutaneous coronary intervention with intracoronary pressure wire guidance. J Am Coll Cardiol 2020;75:2785-99.
- 18. Norgaaard BL, Terkelsen CJ, Mathiassen ON, Grove EL, Botker HE, Parner E, et al. Coronary CT Angiographic and Flow Reserve-Guided Management of Patients with Stable Ischemic Heart Disease. J Am Coll Cardiol 2018;72:2123-34
- 19. Patel MR, Norgaard BL, Fairbairn TA, Nieman K, Akasaka T, Berman DS, et al. 1-Year Impact on Medical Practice and Clinical Outcomes of FFRCT. The ADVANCE Registry. JACC Cardiovasc Imaging 2020;13:97-105.
- 20. Collet C, Onuma Y, Andreini D, Sonck J, Pompilio G, Mustaq S, et al. Coronary computed tomography angiography for heart team decision-making in multivessel coronary artery disease. Eur Heart J 2018; 39:3689-98.


- 21. Krievins D, Zellans E, Erglis A, Zvaigzne L, Lacis A, Jegere S et al. High prevalence of asymptomatic ischemia-producing coronary stenosis in patients with critical limb ischemia. Vascular disease management 2018;15:E96-E101
- 22. Krievins D, Zellans E, Latkovskis G, Erglis A, Zvaigzne L, Kumsars I, et al. Pre-operative diagnosis of silent coronary ischemia may reduce post-operative death and myocardial infarction and improve survival of patients undergoing lower-extremity surgical revascularization. Eur J Vasc Endovasc Surg 2020;60:411-20
- 23. Krievins D, Zellans E, Latkovskis G, Kumsars I, Jegere S, Rumba R, et al. Diagnosis of silent coronary ischemia with selective coronary revascularization may improve two-year survival of patients with critical limb threatening ischemia. J Vasc Surg 2021; doi.org/10.1016/j.jvs.2021.03.059.
- 24. Abbara S, Blanke P, Maroules CD, Cheezum M, Choi AD, Han BK, et al. SCCT guidelines for the performance and acquisition of coronary computed tomographic angiography. J Cardiovasc Comput Tomogr 2016;10(6):435-49.
- 25. Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, et al. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J 2019;40:87-165.
- 26. Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, et al. Standardized End Point Definitions for Coronary Intervention Trials. Circulation 2018;137:2635-2650.
- 27. Latkovskis G, Zellans E, Krievina A, Kumsars I, Jegere S, Erglis A, et al. FFR<sub>CT</sub>-guided revascularization of silent coronary ischemia compared to best medical therapy following lower-extremity revascularization. Interv Cardiol 2021;13,S5:93-102.
- 28. Johnson NP, Toth GG, Lai D, Zhu H, Acar G, Agostoni Pet al. Prognostic value of fractional flow reserve: linking physiologic severity to clinical outcomes. J Am Coll Cardiol 2014;64:1641-54.
- 29. Ciccarelli G, Barbato E, Toth GG, Gahl B, Xaplanteris P, Fournier S et al. Angiography versus hemodynamics to predict the natural history of coronary stenoses: fractional flow reserve versus angiography in multivessel evaluation 2 substudy. Circulation 2018;137:1475-85.
- 30. Dinh K, Gomes ML, Thomas SD, Paravastu SCV, Holden A, Schneider PA, et al. Mortality after paclitaxel-coated device use in patients with chronic limb-threatening ischemia: a systematic review and meta-analysis of randomized controlled trials. J Endovasc Ther 2020;27:175-185.
- 31. Nordanstig J, James S, Andersson M, Andersson M, Danielsson P, Gillgren P, et al. Mortality with paclitaxel-coated devices in 347 peripheral artery disease. N Engl J Med 2020;3832538-46.
- 32. Navarese EP, Lansky AJ, Kereiakes DJ, Kubica J, Gurbel PA, Gorog DA, et al. Cardiac mortality in patients randomised to elective coronary revascularization plus medical therapy or medical therapy alone: a systematic review and meta-analysis. Eur Heart J 2021;00:1-14.

